CLINICAL TRIAL: NCT01850082
Title: CSP #588 - Randomized Endo-Vein Graft Prospective (REGROUP) Trial
Brief Title: Randomized Endo-Vein Graft Prospective
Acronym: REGROUP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 588
Record Dates: First submitted 2013-04-18; First posted 2013-05-09 (Estimated); Results first posted 2021-11-11 (Actual); Last update posted 2021-12-15 (Actual); Status verified 2021-11

CONDITIONS: Coronary Artery Bypass Grafting
Keywords: Coronary artery disease; CABG; Coronary revascularization; Endoscopic vein harvest; Saphenous vein graft; Graft failure
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Endoscopic Vein Harvest (EVH) (Other): An endoscopic vein harvest allows a portion of vein from the inside of the leg to be removed through small incisions. This reduces the length of the incision by several inches. An endoscope, or video camera, is used to view the vein and remove the needed length.
  Interventions: Procedure: Vein Harvesting Procedures
- Open Vein Harvest (OVH) (Other): Open vein harvesting is the traditional method for vein harvesting. It is performed under direct vision using a single long incision or, more commonly, multiple-smaller incisions (referred to as "bridging" technique) along the course of the vein.
  Interventions: Procedure: Vein Harvesting Procedures

INTERVENTIONS:
Procedure: Vein Harvesting Procedures — Open Vein Harvesting is the traditional method of saphenectomy for CABG. It is performed under direct vision using a single long incision or, more commonly, multiple smaller incisions (referred to as "bridging" technique) along the course of the vein. This approach minimizes manipulation and direct trauma to the conduit but is associated with potential for discomfort and leg wound healing complications. Endoscopic Vein Harvesting is a minimally invasive procedure that was developed to eliminate the need for long incisions associated with OVH. EVH reduces the risk of wound infections and other leg wound complications but may be more traumatic to the conduit than OVH.

SUMMARY:
Coronary artery bypass grafting (CABG) is the most common major surgical procedure in the United States with over 300,000 cases performed each year. To restore blood flow to the heart, vascular conduits from another part of the body are procured to create a bypass around critically blocked coronary arteries. The left internal thoracic artery is the conduit of choice for CABG due to its superior long-term patency. However, almost all patients referred for CABG require additional grafts to provide complete revascularization. This necessitates the harvest of other vessels, most commonly the saphenous vein which is used almost ubiquitously in contemporary CABG with an average of two vein grafts per CABG procedure. In the last 10 years, Endoscopic Vein Harvesting (EVH) has been recommended as the preferred method over the traditional open harvesting technique (OVH) because it provides a minimally invasive approach. However, more recent investigations indicate potential for reduced long-term bypass graft patency and worse clinical outcomes with EVH. The long term impact of EVH on clinical outcomes has never been investigated on a large scale using a definitive, adequately powered, prospective Randomized Controlled Trial (RCT) with long-term follow-up.

DETAILED DESCRIPTION:
CSP #588 - REGROUP is a randomized, intent-to-treat, two-arm, parallel design, multicenter study. Cardiac Surgery Programs at Veterans Affairs Medical Centers (VAMC) with expertise in performing both EVH and OVH will be invited to participate in the study. Subjects requiring elective or urgent CABG using cardiopulmonary bypass with use of at least one SVG will be screened for enrollment using established inclusion/exclusion criteria. Enrolled Subjects will be randomized to one of the two arms (EVH or OVH) after an experienced vein harvester is identified and assigned. Intraoperative assessments will be collected and post-operative assessments will be completed 24 hours post-surgery. Additional assessments will be completed at the time of discharge or at the 30-day post-surgery date if the subject is still in the hospital. Assessment of leg wound complications will be completed at the time of discharge and at six-week post-surgery. Telephone follow-ups will occur at three-month interval post-surgery until the participating sites are decommissioned at the end of the trial period (which would be approximately 4.5 years after the site initiations). For long-term MACE outcomes, passive follow up for MACE events using VA databases (CPRS, VASQIP) will be performed centrally by the Study Chair's office for another 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Age years 18 years or older
* Elective or Urgent CABG-only
* Median sternotomy approach
* At least one coronary bypass planned using saphenous vein graft for conduit
* Experienced EVH/OVH harvester available for procedure

Exclusion Criteria:

* Combined valve procedure planned
* Moderate or severe valve disease (see definition of moderate/severe valve)
* Hemodynamically unstable or in cardiogenic shock
* Enrolled in another therapeutic or interventional study
* Off-pump CABG procedure planned
* Limited life expectancy < 1 year
* History of lower extremities venous stripping or ligation
* Inability to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1150 (Actual)
Dates: Start 2013-09-30 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-10-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marco A Zenati, MD MSc, Study Chair — VA Boston Healthcare System Jamaica Plain Campus, Jamaica Plain, MA
Locations (16):
- United States (16):
  - Southern Arizona VA Health Care System, Tucson, AZ, Tucson, Arizona
  - San Francisco VA Medical Center, San Francisco, CA, San Francisco, California
  - North Florida/South Georgia Veterans Health System, Gainesville, FL, Gainesville, Florida
  - Miami VA Healthcare System, Miami, FL, Miami, Florida
  - James A. Haley Veterans' Hospital, Tampa, FL, Tampa, Florida
  - VA Boston Healthcare System Jamaica Plain Campus, Jamaica Plain, MA, Boston, Massachusetts
  - Minneapolis VA Health Care System, Minneapolis, MN, Minneapolis, Minnesota
  - New Mexico VA Health Care System, Albuquerque, NM, Albuquerque, New Mexico
  - Manhattan Campus of the VA NY Harbor Healthcare System, New York, NY, New York, New York
  - Asheville VA Medical Center, Asheville, NC, Asheville, North Carolina
  - Durham VA Medical Center, Durham, NC, Durham, North Carolina
  - Louis Stokes VA Medical Center, Cleveland, OH, Cleveland, Ohio
  - VA Portland Health Care System, Portland, OR, Portland, Oregon
  - VA Pittsburgh Healthcare System University Drive Division, Pittsburgh, PA, Pittsburgh, Pennsylvania
  - Michael E. DeBakey VA Medical Center, Houston, TX, Houston, Texas
  - Clement J. Zablocki VA Medical Center, Milwaukee, WI, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zenati MA, Gaziano JM, Collins JF, Biswas K, Gabany JM, Quin JA, Bitondo JM, Bakaeen FG, Kelly RF, Shroyer AL, Bhatt DL. Choice of vein-harvest technique for coronary artery bypass grafting: rationale and design of the REGROUP trial. Clin Cardiol. 2014 Jun;37(6):325-30. doi: 10.1002/clc.22267. Epub 2014 Mar 14. PMID 24633760
- [Derived] Almassi GH, Quin JA, Stock EM, DeMatt EJ, Biswas K, Hattler B, Tseng E, Zenati MA. Impact of Oral Anticoagulation on Clinical Outcomes in Postoperative Atrial Fibrillation. J Surg Res. 2024 Mar;295:122-130. doi: 10.1016/j.jss.2023.10.016. Epub 2023 Nov 25. PMID 38007859
- [Derived] Gikandi A, Habertheuer A, Stock EM, Hirji S, Kinlay S, Tsao A, Butala N, Biswas K, Zenati MA. Anatomical SYNTAX score and major adverse cardiac events following CABG in the REGROUP trial. J Cardiol. 2024 May;83(5):348-350. doi: 10.1016/j.jjcc.2023.11.003. Epub 2023 Nov 17. No abstract available. PMID 37977259
- [Derived] Wagner TH, Hattler B, Stock EM, Biswas K, Bhatt DL, Bakaeen FG, Gujral K, Zenati MA. Costs of Endoscopic vs Open Vein Harvesting for Coronary Artery Bypass Grafting: A Secondary Analysis of the REGROUP Trial. JAMA Netw Open. 2022 Jun 1;5(6):e2217686. doi: 10.1001/jamanetworkopen.2022.17686. PMID 35727582
- [Derived] Shapeton AD, Leissner KB, Zorca SM, Amirfarzan H, Stock EM, Biswas K, Haime M, Srinivasa V, Quin JA, Zenati MA. Epiaortic Ultrasound for Assessment of Intraluminal Atheroma; Insights from the REGROUP Trial. J Cardiothorac Vasc Anesth. 2020 Mar;34(3):726-732. doi: 10.1053/j.jvca.2019.10.053. Epub 2019 Nov 9. PMID 31787434
- [Derived] Zenati MA, Bhatt DL, Bakaeen FG, Stock EM, Biswas K, Gaziano JM, Kelly RF, Tseng EE, Bitondo J, Quin JA, Almassi GH, Haime M, Hattler B, DeMatt E, Scrymgeour A, Huang GD; REGROUP Trial Investigators. Randomized Trial of Endoscopic or Open Vein-Graft Harvesting for Coronary-Artery Bypass. N Engl J Med. 2019 Jan 10;380(2):132-141. doi: 10.1056/NEJMoa1812390. Epub 2018 Nov 11. PMID 30417737

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Endoscopic Vein Harvest (EVH) | Open Vein Harvest (OVH)
Started | 576 | 574
Completed | 576 | 574
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Endoscopic Vein Harvest (EVH) | Open Vein Harvest (OVH) | Total
Number analyzed (Participants) | 576 | 574 | 1150
Age, Continuous [Mean (Standard Deviation); unit: Years] | 66.2 (6.7) | 66.6 (7.1) | 66.4 (6.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 7
  Male | 572 | 571 | 1143
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaskan Native | 4 | 2 | 6
  Asian or Pacific Islander | 6 | 4 | 10
  Black, not of Hispanic origin | 41 | 50 | 91
  Hispanic | 31 | 31 | 62
  , not of Hispanic origin | 490 | 484 | 974
  Other | 3 | 3 | 6
  Missing | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Incidence of First MACE During Active Follow-up Period.
Description: Incidence of first MACE estimated via Kaplan Meier survival analysis (MACE defined as death from any cause, repeat revascularization, myocardial infarction) during the active follow-up period.
Time Frame: Varying timeframe for each participant with a minimum of 1 year and a maximum 4.5 Years
Population: Events captured during the active follow-up phase of the trial (minimum of 1 year and up to 4.5 years) were included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Endoscopic Vein Harvest (EVH) | Open Vein Harvest (OVH)
Number analyzed (Participants) | 576 | 574
Participants | 80 | 89
Statistical Analysis 1: Comparison: Endoscopic Vein Harvest (EVH); Test type: Superiority; p = 0.47, Regression, Cox; Hazard Ratio (HR) = 1.12, 95% CI 2-sided [0.83 to 1.51]

2. Secondary Outcome: MACE at One Year.
Description: Proportion of patients with MACE (death from any cause, repeat revascularization, myocardial infarction) at one year postoperatively.
Time Frame: 1 year
Population: Participants with a minimum of 1 year follow-up or who died within one year.
Measure: Count of Participants; unit: Participants
Arm/Group | Endoscopic Vein Harvest (EVH) | Open Vein Harvest (OVH)
Number analyzed (Participants) | 571 | 570
Participants | 45 | 47
Statistical Analysis 1: Comparison: Endoscopic Vein Harvest (EVH) vs Open Vein Harvest (OVH); Test type: Superiority; p = 0.821, Chi-squared

3. Secondary Outcome: MACE at Three Years.
Description: Proportion of patients with MACE (death from any cause, repeat revascularization, myocardial infarction) at three years postoperatively.
Time Frame: 3 years
Population: Participants with a minimum of 3 years follow-up or died prior to 3 years.
Measure: Count of Participants; unit: Participants
Arm/Group | Endoscopic Vein Harvest (EVH) | Open Vein Harvest (OVH)
Number analyzed (Participants) | 568 | 568
Participants | 90 | 90
Statistical Analysis 1: Comparison: Endoscopic Vein Harvest (EVH) vs Open Vein Harvest (OVH); Test type: Superiority; p > 0.99, Chi-squared

4. Secondary Outcome: Incidence of First MACE Over the Entire Follow-up Period (Active and Passive).
Description: Incidence of first MACE estimated via Kaplan Meier survival analysis (MACE defined as death from any cause, repeat revascularization, myocardial infarction) during the entire follow-up period (active and passive).
Time Frame: Varying timeframe for each participant with a minimum of 3 years and a maximum of 6.5 years
Population: Events captured throughout active and passive follow-up are included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Endoscopic Vein Harvest (EVH) | Open Vein Harvest (OVH)
Number analyzed (Participants) | 576 | 574
Participants | 126 | 135
Statistical Analysis 1: Comparison: Endoscopic Vein Harvest (EVH) vs Open Vein Harvest (OVH); Test type: Superiority; p = 0.517, Regression, Cox; Hazard Ratio (HR) = 0.923, 95% CI 2-sided [0.724 to 1.176]

ADVERSE EVENTS:
Time Frame: Participant adverse event data collection stopped at the end of active follow-up. All participants had a minimum of 1 year of SAE reporting with a maximum duration of 4 years 7 months, depending on participants' time of termination from active follow-up. However, all cause mortality was collected through passive follow-up (6.5 years).
Description: Only Serious Adverse Events were collected. Collection of SAE's occurred through routine inquiry by Site Investigator every 3 months at study visits/phone call assessments.
Arm/Group | Endoscopic Vein Harvest (EVH) | Open Vein Harvest (OVH)
All-Cause Mortality (participants affected / at risk) | 69/576 | 76/574
Serious Adverse Events (participants affected / at risk) | 366/576 | 359/574
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Endoscopic Vein Harvest (EVH) (N=576) | Open Vein Harvest (OVH) (N=574)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Coagulopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Haemorrhagic disorder (Blood and lymphatic system disorders) | 0 (0) | 0 (0)
Heparin-induced thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Immune thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Splenic haematoma (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Acute coronary syndrome (Cardiac disorders) | 2 (2) | 1 (1)
Acute left ventricular failure (Cardiac disorders) | 2 (2) | 0 (0)
Angina pectoris (Cardiac disorders) | 8 (8) | 8 (11)
Angina unstable (Cardiac disorders) | 3 (3) | 6 (7)
Aortic valve stenosis (Cardiac disorders) | 1 (1) | 0 (0)
Arrhythmia (Cardiac disorders) | 0 (0) | 2 (2)
Arteriosclerosis coronary artery (Cardiac disorders) | 3 (3) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 25 (30) | 31 (36)
Atrial flutter (Cardiac disorders) | 15 (16) | 3 (3)
Atrial tachycardia (Cardiac disorders) | 2 (2) | 0 (0)
Atrioventricular block (Cardiac disorders) | 0 (0) | 1 (1)
Atrioventricular block complete (Cardiac disorders) | 4 (4) | 3 (3)
Atrioventricular block first degree (Cardiac disorders) | 0 (0) | 1 (1)
Atrioventricular block second degree (Cardiac disorders) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 3 (3) | 4 (5)
Cardiac arrest (Cardiac disorders) | 3 (3) | 2 (2)
Cardiac failure (Cardiac disorders) | 6 (6) | 9 (12)
Cardiac failure acute (Cardiac disorders) | 4 (4) | 4 (5)
Cardiac failure congestive (Cardiac disorders) | 41 (53) | 25 (50)
Cardiac perforation (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac tamponade (Cardiac disorders) | 0 (0) | 1 (1)
Cardiogenic shock (Cardiac disorders) | 2 (2) | 2 (2)
Cardiomyopathy (Cardiac disorders) | 2 (2) | 0 (0)
Cor pulmonale (Cardiac disorders) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 23 (26) | 30 (34)
Coronary artery occlusion (Cardiac disorders) | 2 (2) | 7 (7)
Coronary artery stenosis (Cardiac disorders) | 8 (8) | 5 (6)
Coronary ostial stenosis (Cardiac disorders) | 0 (0) | 1 (1)
Defect conduction intraventricular (Cardiac disorders) | 1 (1) | 1 (1)
Intracardiac thrombus (Cardiac disorders) | 1 (1) | 0 (0)
Ischaemic cardiomyopathy (Cardiac disorders) | 2 (2) | 0 (0)
Left ventricular dysfunction (Cardiac disorders) | 0 (0) | 1 (1)
Left ventricular failure (Cardiac disorders) | 1 (1) | 1 (1)
Mitral valve incompetence (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 27 (28) | 30 (34)
Myocardial ischaemia (Cardiac disorders) | 1 (1) | 2 (2)
Nodal rhythm (Cardiac disorders) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 3 (3) | 0 (0)
Papillary muscle rupture (Cardiac disorders) | 1 (1) | 0 (0)
Pericardial effusion (Cardiac disorders) | 5 (5) | 5 (9)
Pericardial haemorrhage (Cardiac disorders) | 2 (2) | 0 (0)
Pericarditis (Cardiac disorders) | 1 (1) | 2 (3)
Pericarditis uraemic (Cardiac disorders) | 0 (0) | 1 (1)
Pulseless electrical activity (Cardiac disorders) | 0 (0) | 1 (1)
Right ventricular failure (Cardiac disorders) | 0 (0) | 1 (1)
Sinus arrest (Cardiac disorders) | 0 (0) | 1 (1)
Sinus node dysfunction (Cardiac disorders) | 3 (3) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 2 (2)
Tachycardia (Cardiac disorders) | 2 (2) | 0 (0)
Ventricular arrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular asystole (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular extrasystoles (Cardiac disorders) | 2 (2) | 2 (2)
Ventricular fibrillation (Cardiac disorders) | 3 (4) | 4 (4)
Ventricular tachycardia (Cardiac disorders) | 4 (5) | 4 (4)
Meniere's disease (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 2 (2)
Adrenocortical insufficiency acute (Endocrine disorders) | 0 (0) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 1 (1)
Thyroid disorder (Endocrine disorders) | 0 (0) | 1 (1)
Diplopia (Eye disorders) | 1 (1) | 0 (0)
Endocrine ophthalmopathy (Eye disorders) | 0 (0) | 1 (1)
Optic ischaemic neuropathy (Eye disorders) | 1 (1) | 0 (0)
Retinal detachment (Eye disorders) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal hernia (Gastrointestinal disorders) | 0 (0) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 2 (2)
Abdominal wall haematoma (Gastrointestinal disorders) | 1 (1) | 0 (0)
Anal stenosis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 4 (4)
Colitis ischaemic (Gastrointestinal disorders) | 1 (2) | 1 (1)
Colonic pseudo-obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 3 (3)
Dieulafoy's vascular malformation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diverticulum (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 0 (0) | 1 (1)
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1 (1) | 2 (2)
Dysphagia (Gastrointestinal disorders) | 2 (2) | 3 (3)
Enteritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 1 (2)
Enterocutaneous fistula (Gastrointestinal disorders) | 1 (1) | 0 (0)
Epiploic appendagitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Food poisoning (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 2 (2) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastritis erosive (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 4 (4) | 2 (2)
Gastrointestinal polyp haemorrhage (Gastrointestinal disorders) | 2 (2) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 (2) | 5 (5)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 (1) | 2 (2)
Ileus (Gastrointestinal disorders) | 1 (1) | 2 (2)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Large intestinal stenosis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Large intestinal ulcer haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Large intestine perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mallory-Weiss syndrome (Gastrointestinal disorders) | 0 (0) | 1 (1)
Melaena (Gastrointestinal disorders) | 0 (0) | 1 (1)
Obstruction gastric (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oesophageal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oesophageal stenosis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oesophageal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oral disorder (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (3) | 2 (2)
Pancreatitis acute (Gastrointestinal disorders) | 3 (3) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1)
Salivary gland cyst (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Umbilical hernia (Gastrointestinal disorders) | 0 (0) | 2 (2)
Varices oesophageal (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 3 (3) | 2 (2)
Adverse drug reaction (General disorders) | 0 (0) | 3 (4)
Asthenia (General disorders) | 3 (3) | 2 (2)
Brain death (General disorders) | 1 (1) | 0 (0)
Cardiac death (General disorders) | 0 (0) | 1 (1)
Catheter site haematoma (General disorders) | 0 (0) | 1 (1)
Chest discomfort (General disorders) | 4 (4) | 1 (1)
Chest pain (General disorders) | 23 (24) | 28 (34)
Complication associated with device (General disorders) | 2 (2) | 0 (0)
Complication of device removal (General disorders) | 1 (1) | 0 (0)
Death (General disorders) | 4 (4) | 3 (3)
Device related thrombosis (General disorders) | 0 (0) | 1 (1)
Drug withdrawal syndrome (General disorders) | 0 (0) | 1 (1)
Impaired healing (General disorders) | 0 (0) | 3 (3)
Ischaemic ulcer (General disorders) | 1 (1) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 11 (12) | 13 (13)
Pacemaker generated arrhythmia (General disorders) | 1 (1) | 1 (1)
Peripheral swelling (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 3 (3) | 0 (0)
Submandibular mass (General disorders) | 0 (0) | 1 (1)
Sudden cardiac death (General disorders) | 0 (0) | 2 (2)
Systemic inflammatory response syndrome (General disorders) | 1 (1) | 1 (1)
Vascular stent thrombosis (General disorders) | 0 (0) | 1 (1)
Bile duct obstruction (Hepatobiliary disorders) | 0 (0) | 1 (1)
Bile duct stone (Hepatobiliary disorders) | 1 (1) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 2 (2) | 3 (3)
Cholecystitis acute (Hepatobiliary disorders) | 5 (6) | 3 (3)
Cholelithiasis (Hepatobiliary disorders) | 2 (2) | 3 (3)
Drug-induced liver injury (Hepatobiliary disorders) | 1 (1) | 0 (0)
Gallbladder disorder (Hepatobiliary disorders) | 0 (0) | 1 (1)
Gallbladder perforation (Hepatobiliary disorders) | 0 (0) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 1 (1) | 1 (1)
Abdominal wall abscess (Infections and infestations) | 1 (1) | 0 (0)
Abscess limb (Infections and infestations) | 1 (1) | 0 (0)
Abscess neck (Infections and infestations) | 1 (1) | 0 (0)
Acute sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Anal abscess (Infections and infestations) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 2 (2) | 1 (1)
Arthritis bacterial (Infections and infestations) | 1 (1) | 0 (0)
Bacteraemia (Infections and infestations) | 2 (2) | 1 (1)
Bronchitis (Infections and infestations) | 4 (4) | 2 (2)
Cellulitis (Infections and infestations) | 12 (15) | 11 (13)
Cellulitis staphylococcal (Infections and infestations) | 0 (0) | 1 (1)
Clostridium difficile colitis (Infections and infestations) | 1 (1) | 2 (2)
Clostridium difficile infection (Infections and infestations) | 0 (0) | 3 (3)
Colonic abscess (Infections and infestations) | 1 (1) | 0 (0)
Device related infection (Infections and infestations) | 0 (0) | 1 (1)
Diabetic foot infection (Infections and infestations) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 2 (2) | 2 (2)
Endocarditis (Infections and infestations) | 1 (1) | 1 (1)
Enteritis infectious (Infections and infestations) | 0 (0) | 1 (1)
Enterobacter sepsis (Infections and infestations) | 0 (0) | 1 (1)
Enterococcal bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Epididymitis (Infections and infestations) | 0 (0) | 1 (1)
Epiglottitis (Infections and infestations) | 1 (1) | 0 (0)
Gangrene (Infections and infestations) | 2 (6) | 1 (1)
Gastroenteritis (Infections and infestations) | 4 (4) | 4 (4)
Haematoma infection (Infections and infestations) | 1 (1) | 0 (0)
Haemophilus infection (Infections and infestations) | 0 (0) | 1 (1)
Implant site infection (Infections and infestations) | 2 (2) | 0 (0)
Incision site cellulitis (Infections and infestations) | 2 (2) | 4 (4)
Incision site infection (Infections and infestations) | 0 (0) | 2 (2)
Infected skin ulcer (Infections and infestations) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 3 (3) | 2 (2)
Localised infection (Infections and infestations) | 7 (7) | 15 (15)
Mediastinitis (Infections and infestations) | 2 (2) | 0 (0)
Medical device site infection (Infections and infestations) | 0 (0) | 1 (1)
Meningitis (Infections and infestations) | 0 (0) | 1 (2)
Osteomyelitis (Infections and infestations) | 5 (5) | 4 (8)
Perirectal abscess (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 39 (51) | 36 (40)
Post procedural pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Postoperative wound infection (Infections and infestations) | 19 (27) | 18 (20)
Sepsis (Infections and infestations) | 4 (4) | 2 (2)
Septic shock (Infections and infestations) | 1 (1) | 1 (1)
Streptococcal infection (Infections and infestations) | 1 (1) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 1 (1) | 0 (0)
Subdural empyema (Infections and infestations) | 0 (0) | 1 (1)
Tracheobronchitis (Infections and infestations) | 3 (3) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 2 (2)
Urinary tract infection (Infections and infestations) | 5 (5) | 10 (10)
Urosepsis (Infections and infestations) | 0 (0) | 1 (1)
Viral infection (Infections and infestations) | 1 (1) | 1 (1)
Wound abscess (Infections and infestations) | 1 (1) | 0 (0)
Wound infection (Infections and infestations) | 1 (1) | 0 (0)
Agitation postoperative (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Alcohol poisoning (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Anaemia postoperative (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Arteriovenous fistula site haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Brachial plexus injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Coronary vascular graft occlusion (Injury, poisoning and procedural complications) | 5 (6) | 3 (3)
Deep vein thrombosis postoperative (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Endotracheal intubation complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Extradural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Facial bones fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 3 (3) | 1 (1)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Gastrointestinal injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Graft haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Haemodialysis-induced symptom (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Incision site complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Incision site haematoma (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Incision site haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Incision site pain (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Lower limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Mental status changes postoperative (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Multiple fractures (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (2)
Pelvic fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Perirenal haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Peritoneal dialysis complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post procedural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural haematuria (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 6 (6) | 4 (4)
Post procedural myocardial infarction (Injury, poisoning and procedural complications) | 1 (1) | 4 (4)
Post procedural swelling (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Postoperative ileus (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Postoperative respiratory distress (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Postoperative respiratory failure (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Postoperative thoracic procedure complication (Injury, poisoning and procedural complications) | 3 (3) | 1 (1)
Postoperative wound complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Procedural complication (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Procedural hypotension (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Procedural pneumothorax (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Procedural site reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Radiation dysphagia (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Radiation proctitis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Scrotal haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Seroma (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Spinal cord injury (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Subarachnoid haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (2) | 2 (2)
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Traumatic fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (2)
Vascular graft occlusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vascular graft stenosis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vasoplegia syndrome (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wound (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wound dehiscence (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Anticoagulation drug level above therapeutic (Investigations) | 1 (1) | 0 (0)
Arthroscopy (Investigations) | 0 (0) | 1 (1)
Blood potassium decreased (Investigations) | 0 (0) | 1 (1)
Electrocardiogram QT prolonged (Investigations) | 0 (0) | 1 (1)
Electroencephalogram (Investigations) | 1 (1) | 0 (0)
Influenza B virus test positive (Investigations) | 0 (0) | 1 (1)
International normalised ratio increased (Investigations) | 0 (0) | 2 (2)
Medical observation (Investigations) | 1 (1) | 0 (0)
Oxygen consumption increased (Investigations) | 1 (1) | 0 (0)
Oxygen saturation decreased (Investigations) | 1 (1) | 0 (0)
Transaminases increased (Investigations) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 9 (9)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 (1) | 2 (3)
Failure to thrive (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Fluid overload (Metabolism and nutrition disorders) | 2 (4) | 5 (6)
Fluid retention (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Gout (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 3 (3) | 1 (1)
Hyperglycaemic hyperosmolar nonketotic syndrome (Metabolism and nutrition disorders) | 0 (0) | 1 (3)
Hyperkalaemia (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 6 (6)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypovolaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Costochondritis (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1)
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 7 (9) | 12 (12)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Myopathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Myositis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 9 (10) | 10 (10)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Vertebral foraminal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (3) | 0 (0)
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0)
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Carcinoid tumour pulmonary (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2)
Clear cell renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (3) | 1 (4)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung adenocarcinoma stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 3 (3)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 3 (3)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Non-Hodgkin's lymphoma stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Non-small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Oesophageal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 2 (3)
Oropharyngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Pituitary tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (3)
Small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (3)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0)
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Tumour necrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Amyotrophic lateral sclerosis (Nervous system disorders) | 1 (2) | 0 (0)
Autonomic nervous system imbalance (Nervous system disorders) | 0 (0) | 1 (1)
Basal ganglia haemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Brain hypoxia (Nervous system disorders) | 0 (0) | 1 (1)
Carotid artery stenosis (Nervous system disorders) | 6 (7) | 4 (5)
Carotid artery thrombosis (Nervous system disorders) | 0 (0) | 1 (1)
Cerebellar infarction (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 1 (1) | 1 (1)
Cerebral infarction (Nervous system disorders) | 2 (2) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 17 (22) | 20 (23)
Cervical myelopathy (Nervous system disorders) | 1 (1) | 1 (1)
Clonus (Nervous system disorders) | 1 (1) | 0 (0)
Cognitive disorder (Nervous system disorders) | 0 (0) | 1 (1)
Dementia (Nervous system disorders) | 1 (1) | 2 (2)
Dementia Alzheimer's type (Nervous system disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 4 (4) | 0 (0)
Dizziness postural (Nervous system disorders) | 0 (0) | 1 (1)
Dyskinesia (Nervous system disorders) | 0 (0) | 1 (1)
Embolic stroke (Nervous system disorders) | 1 (1) | 0 (0)
Encephalopathy (Nervous system disorders) | 2 (2) | 1 (1)
Epilepsy (Nervous system disorders) | 1 (1) | 0 (0)
Generalised tonic-clonic seizure (Nervous system disorders) | 1 (1) | 1 (1)
Haemorrhagic cerebral infarction (Nervous system disorders) | 0 (0) | 1 (1)
Haemorrhagic stroke (Nervous system disorders) | 0 (0) | 1 (1)
Hemiparesis (Nervous system disorders) | 0 (0) | 1 (1)
Horner's syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Intensive care unit acquired weakness (Nervous system disorders) | 0 (0) | 1 (1)
Loss of consciousness (Nervous system disorders) | 0 (0) | 1 (1)
Lumbar radiculopathy (Nervous system disorders) | 2 (2) | 0 (0)
Migraine (Nervous system disorders) | 1 (1) | 1 (1)
Monoparesis (Nervous system disorders) | 0 (0) | 1 (1)
Neuralgia (Nervous system disorders) | 1 (1) | 0 (0)
Neuroleptic malignant syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 3 (3) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Poor quality sleep (Nervous system disorders) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 3 (3) | 1 (1)
Seizure (Nervous system disorders) | 2 (3) | 4 (4)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 7 (8) | 3 (3)
Transient ischaemic attack (Nervous system disorders) | 6 (6) | 3 (3)
Vertebral artery thrombosis (Nervous system disorders) | 0 (0) | 1 (1)
Device dislocation (Product Issues) | 1 (2) | 1 (1)
Device failure (Product Issues) | 1 (1) | 0 (0)
Device kink (Product Issues) | 1 (1) | 0 (0)
Device malfunction (Product Issues) | 1 (1) | 0 (0)
Aggression (Psychiatric disorders) | 2 (2) | 1 (1)
Alcohol withdrawal syndrome (Psychiatric disorders) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 3 (4) | 2 (3)
Bipolar disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Conversion disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Delirium (Psychiatric disorders) | 2 (2) | 2 (2)
Delirium tremens (Psychiatric disorders) | 1 (1) | 1 (1)
Depression (Psychiatric disorders) | 2 (2) | 0 (0)
Drug use disorder (Psychiatric disorders) | 1 (1) | 1 (1)
Homicidal ideation (Psychiatric disorders) | 1 (1) | 1 (1)
Major depression (Psychiatric disorders) | 0 (0) | 1 (1)
Mental status changes (Psychiatric disorders) | 2 (2) | 2 (2)
Panic attack (Psychiatric disorders) | 1 (1) | 0 (0)
Stress (Psychiatric disorders) | 0 (0) | 1 (1)
Substance use disorder (Psychiatric disorders) | 1 (1) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 5 (6) | 5 (11)
Suicide attempt (Psychiatric disorders) | 1 (1) | 0 (0)
Violence-related symptom (Psychiatric disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 16 (19) | 13 (17)
Chronic kidney disease (Renal and urinary disorders) | 3 (3) | 1 (1)
Diabetic nephropathy (Renal and urinary disorders) | 0 (0) | 1 (1)
End stage renal disease (Renal and urinary disorders) | 1 (1) | 6 (7)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (2)
Nephrolithiasis (Renal and urinary disorders) | 2 (2) | 1 (1)
Nephrotic syndrome (Renal and urinary disorders) | 0 (0) | 1 (2)
Polyuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal artery stenosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 0 (0) | 3 (3)
Renal mass (Renal and urinary disorders) | 1 (1) | 1 (1)
Renal tubular necrosis (Renal and urinary disorders) | 2 (2) | 0 (0)
Ureterolithiasis (Renal and urinary disorders) | 1 (1) | 1 (1)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 1 (1)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 2 (2) | 5 (5)
Erectile dysfunction (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Bronchial secretion retention (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Choking (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 10 (17) | 13 (18)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Diaphragmatic paralysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 4 (4)
Mediastinal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 25 (27) | 17 (23)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (4)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2)
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 9 (10) | 9 (9)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 11 (11)
Thoracic haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Angioedema (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Cold sweat (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Diabetic foot (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 2 (3) | 3 (3)
Homeless (Social circumstances) | 1 (1) | 1 (1)
Abdominal panniculectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Ankle arthroplasty (Surgical and medical procedures) | 1 (1) | 0 (0)
Arteriovenous fistula operation (Surgical and medical procedures) | 0 (0) | 1 (1)
Arteriovenous graft (Surgical and medical procedures) | 0 (0) | 1 (1)
Bladder neoplasm surgery (Surgical and medical procedures) | 0 (0) | 3 (4)
Cardiac pacemaker replacement (Surgical and medical procedures) | 1 (1) | 0 (0)
Cardioversion (Surgical and medical procedures) | 1 (1) | 1 (1)
Chemotherapy (Surgical and medical procedures) | 0 (0) | 1 (1)
Cholecystectomy (Surgical and medical procedures) | 1 (1) | 1 (1)
Coronary revascularisation (Surgical and medical procedures) | 0 (0) | 1 (1)
Debridement (Surgical and medical procedures) | 2 (2) | 2 (2)
Dialysis device insertion (Surgical and medical procedures) | 0 (0) | 1 (1)
Drug rehabilitation (Surgical and medical procedures) | 0 (0) | 1 (2)
Elective procedure (Surgical and medical procedures) | 1 (1) | 0 (0)
Gastrointestinal tube insertion (Surgical and medical procedures) | 1 (1) | 0 (0)
Hip arthroplasty (Surgical and medical procedures) | 0 (0) | 5 (5)
Incisional drainage (Surgical and medical procedures) | 1 (1) | 2 (2)
Intervertebral disc operation (Surgical and medical procedures) | 1 (1) | 0 (0)
Knee arthroplasty (Surgical and medical procedures) | 0 (0) | 2 (2)
Medical device removal (Surgical and medical procedures) | 1 (1) | 0 (0)
Metabolic surgery (Surgical and medical procedures) | 1 (1) | 0 (0)
Multiple drug therapy (Surgical and medical procedures) | 1 (1) | 0 (0)
Nephrectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Pancreatic stent placement (Surgical and medical procedures) | 1 (1) | 0 (0)
Parotidectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Peripheral artery bypass (Surgical and medical procedures) | 0 (0) | 1 (1)
Renal transplant (Surgical and medical procedures) | 0 (0) | 1 (1)
Shoulder arthroplasty (Surgical and medical procedures) | 1 (1) | 0 (0)
Spinal fusion surgery (Surgical and medical procedures) | 1 (1) | 0 (0)
Spinal laminectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Spinal operation (Surgical and medical procedures) | 0 (0) | 1 (1)
Sternal wiring (Surgical and medical procedures) | 1 (1) | 0 (0)
Suture removal (Surgical and medical procedures) | 0 (0) | 1 (1)
Wound drainage (Surgical and medical procedures) | 0 (0) | 3 (3)
Aneurysm (Vascular disorders) | 1 (1) | 0 (0)
Aortic aneurysm (Vascular disorders) | 2 (2) | 6 (6)
Aortic dissection (Vascular disorders) | 0 (0) | 3 (3)
Arteriosclerosis (Vascular disorders) | 0 (0) | 2 (2)
Deep vein thrombosis (Vascular disorders) | 5 (6) | 8 (8)
Distributive shock (Vascular disorders) | 0 (0) | 1 (1)
Essential hypertension (Vascular disorders) | 1 (1) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 1 (1)
Haemodynamic instability (Vascular disorders) | 1 (1) | 2 (2)
Hypertension (Vascular disorders) | 1 (1) | 4 (4)
Hypertensive crisis (Vascular disorders) | 1 (1) | 2 (2)
Hypertensive emergency (Vascular disorders) | 2 (2) | 1 (2)
Hypotension (Vascular disorders) | 7 (7) | 7 (7)
Iliac artery occlusion (Vascular disorders) | 0 (0) | 1 (1)
Ischaemia (Vascular disorders) | 0 (0) | 1 (1)
Jugular vein thrombosis (Vascular disorders) | 2 (2) | 1 (1)
Microembolism (Vascular disorders) | 1 (1) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 4 (4) | 5 (6)
Peripheral arterial occlusive disease (Vascular disorders) | 3 (3) | 4 (4)
Peripheral artery aneurysm (Vascular disorders) | 1 (1) | 1 (2)
Peripheral embolism (Vascular disorders) | 0 (0) | 1 (1)
Peripheral ischaemia (Vascular disorders) | 2 (3) | 3 (3)
Peripheral vascular disorder (Vascular disorders) | 2 (3) | 1 (1)
Peripheral venous disease (Vascular disorders) | 0 (0) | 1 (1)
Steal syndrome (Vascular disorders) | 1 (1) | 1 (2)
Subclavian vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Thrombophlebitis superficial (Vascular disorders) | 0 (0) | 1 (1)
Thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Vasculitis (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2013-10-01): https://cdn.clinicaltrials.gov/large-docs/82/NCT01850082/Prot_000.pdf
  • Statistical Analysis Plan (2018-08-30): https://cdn.clinicaltrials.gov/large-docs/82/NCT01850082/SAP_001.pdf